CLINICAL TRIAL: NCT04384042
Title: Olfactory and Gustatory Disturbances as a Clinical Presentation of Coronavirus Disease 2019 (COVID-19) Infection in Malaysia - A Nationwide Multicentre Case-Control Study
Brief Title: Malaysian COVID-19 Anosmia Study (Phase 2) - A Nationwide Multicentre Case-Control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Sultanah Bahiyah (Other Government)
Collaborators: Hospital Tuanku Fauziah, Kangar, Perlis (Unknown); Penang Hospital, Malaysia (Other Government); Hospital Raja Permaisuri Bainun (Other Government); Hospital Sungai Buloh, Selangor (Unknown); Kuala Lumpur General Hospital (Other Government); Hospital Tuanku Jaafar, Seremban, Negeri Sembilan (Unknown); Hospital Melaka, Melaka (Unknown); Hospital Enche Besar Hajjah Khalsom, Kluang, Johor (Unknown); Hospital Raja Perempuan Zainab II, Kota Bahru, Kelantan (Unknown); Hospital Sultanah Nur Zahirah, Kuala Terengganu (Other Government); Hospital Tengku Ampuan Afzan, Kuantan, Pahang (Unknown); Sarawak General Hospital (Other); Hospital Queen Elizabeth, Malaysia (Other Government)
Responsible Party: Principal Investigator, Siti Sabzah bt Mohd Hashim, MD, MS (ORL-HNS), Head of Otorhinolaryngology Service, Ministry of Health, Malaysia & Senior Consultant Otorhinolaryngologist, Hospital Sultanah Bahiyah
Other Study IDs: MCO-002; NMRR-20-934-54803 (Other: National Medical Research Register (NMRR), Malaysia)
Record Dates: First submitted 2020-05-10; First posted 2020-05-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: SARS-CoV Infection; COVID-19; Anosmia; Dysgeusia
Keywords: Cross-sectional study; Prevalence; Otorhinolaryngology; Infectious Diseases; Anosmia; Dysgeusia; Olfactory Disorders; Taste Disorders; COVID-19; SARS-CoV-2; Coronavirus 2019
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Anosmia; Dysgeusia; Communicable Diseases; Taste Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malaysian COVID-19 Cohort (Cases): A cohort of COVID-19 positive patients will be recruited from participating Malaysian Ministry of Health-designated COVID-19 treating hospitals across the country.
  Interventions: Other: Patient-Reported Online Questionnaire on Olfactory & Taste Disturbances
- Healthy Volunteers (Controls): A cohort of age and sex-matched healthy volunteers will be recruited from participating Malaysian Ministry of Health-designated COVID-19 treating hospitals across the country.
  Interventions: Other: Patient-Reported Online Questionnaire on Olfactory & Taste Disturbances

INTERVENTIONS:
Other: Patient-Reported Online Questionnaire on Olfactory & Taste Disturbances — This is an online patient-reported questionnaire that examines the presence or absence of olfactory and taste disturbances, the onset of olfactory and taste disturbances in relation to other COVID-19 symptoms, and the temporal evolution of the severity of olfactory and taste disturbances. The occurrence of ear symptoms in COVID-19 infection will also be evaluated in this questionnaire as a secondary outcome. The questionnaire will also have questions relating to the patient's underlying health conditions, risk factors for COVID-19 infection, and demographics.

SUMMARY:
The Malaysian COVID-19 Anosmia Study is a nationwide multicentre observational study to investigate the prevalence and characteristics of olfactory and gustatory/taste disturbances in COVID-19 infection in Malaysia, and to evaluate the predictive value of screening for these symptoms in COVID-19 infection.

This study consists of two phases: the first phase is a cross-sectional study and the second phase is a case-control study. The case-control study is described here (the cross-sectional study is described in a separate ClinicalTrials.gov record).

DETAILED DESCRIPTION:
The world is currently in the midst of the Coronavirus 2019 (COVID-19) pandemic that is caused by a novel coronavirus, Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). According to published cohort studies on COVID-29 infected patients, the most prevalent symptoms consist of fever, dry cough, dyspnoea, sputum production, myalgia, arthralgia, headache, diarrhoea, and sore throat. Recently, there have been concerns of significant viral transmission through asymptomatic, pre-symptomatic or even mildly symptomatic patients.

There is increasing anecdotal evidence from patients and healthcare professionals highlighting isolated loss of sense of smell (anosmia) and taste disturbances (dysgeusia) as atypical symptoms of COVID-19 infection in otherwise asymptomatic patients. In parallel, expert statements from the British Association of Otorhinolaryngology-Head & Neck Surgery (ENT UK), British Rhinological Society, and the American Association of Otolaryngology-Head & Neck Surgery (AAO-HNS) have suggested that olfactory and taste disturbances could be a clinical feature of COVID-19 infection.

Rapidly emerging evidence from Europe, the United Kingdom and the United States have found olfactory and taste disturbances to be highly prevalent in patients diagnosed with COVID-19. In contrast, there is currently limited evidence from Asia on the prevalence of these symptoms in COVID-19 infection. Additionally, there is also limited evidence on the predictive value of screening for olfactory and taste disturbance in COVID-19 patients with subclinical symptoms.

The aim of this case-control study is to study the predictive value of screening for olfactory and taste disturbance in patients with COVID-19 infection in Malaysia. The cases will be selected from the cohort of COVID-19 positive patients recruited from participating Malaysian Ministry of Health-designated COVID-19 treating hospitals across the country (from Phase 1 of the Malaysian COVID-19 Anosmia Study). Controls will be recruited from healthy volunteers who will will answer the an online questionnaire to evaluate and characterise their olfactory and taste symptoms. This is the same questionnaire that is answered by the COVID-19 patients in case cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years old
2. For Cases: Laboratory confirmed COVID-19 infection [Reverse Transcription Polymerase Chain Reaction (RT-PCR)]
3. Patients clinically able to answer the questionnaire

Exclusion Criteria:

1. Patients with olfactory or taste/gustatory disorders before the COVID-19 epidemic
2. For Cases: Patients without a laboratory-confirmed COVID-19 diagnosis
3. For Cases: Patients in intensive care unit at the time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study population will draw subjects from the cohort in Phase 1 of the Malaysian COVID-19 Anosmia Study (Nationwide Multicentre Cross-Sectional Study) as cases. These cases will comprise adult patients with laboratory-confirmed COVID-19 infection from participating Malaysian hospital sites in this study, since the arrival of COVID-19 infection in Malaysia (January 2020) until present time.
  The control subjects will be age and sex-matched healthy volunteers recruited from participating hospital sites in this study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of olfactory and taste disturbances in study participants | 2 weeks prior to answering questionnaire/ prior to diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked regarding whether they experienced symptoms of olfactory and/or taste disturbances
Adjusted odds ratio of olfactory & taste disturbances in COVID-19 infection | 2 weeks prior to answering questionnaire/ prior to diagnosis of COVID-19 infection
  The relationship between case & control status and each exposure variable will be estimated by odds ratios and their 95% confidence intervals using conditional logistic regression models.

SECONDARY OUTCOMES:
Clinical manifestations of study participants | 2 weeks prior to answering questionnaire/ prior to diagnosis of COVID-19 infection
  In the patient-reported online questionnaire, subjects will be asked regarding other symptoms they experienced when they were diagnosed with COVID-19/within the past 2 weeks of answering the questionnaire (e.g. headache, nasal congestion, fever, chills, cough, dyspnoea, gastrointestinal symptoms, eye & ear symptoms)
Other pre-existing health conditions | Baseline
  In the patient-reported online questionnaire, subjects will be asked regarding their pre-existing health conditions (for example, obesity, diabetes, hypertension, cardiac conditions, previous head trauma, chronic rhinosinusitis, etc.)
Positive predictive value (PPV) of olfactory and taste disturbances in predicting diagnosis of COVID-19 infection | Baseline
  PPV reflects the probability that the presence of olfactory and taste disturbances will have a positive diagnosis of COVID-19. This is derived from dividing the number of patients with olfactory & taste disturbances with COVID-19 infection over the total number of patients with olfactory and taste disturbances, and multiplying by 100%
Negative predictive value (NPV) of olfactory and taste disturbances in predicting absence of COVID-19 infection | Baseline
  NPV reflects the probability that the absence of olfactory and taste disturbances will have a negative diagnosis of COVID-19. This is derived from dividing the number of patients without olfactory & taste disturbances and without COVID-19 infection over the total number of patients with no olfactory and taste disturbances, and multiplying by 100%
Sensitivity of olfactory and taste disturbances in predicting COVID-19 infection | Baseline
  The percentage of true positives, i.e. the proportion of patients with olfactory and taste disorders with COVID-19 infection. This can be calculated by dividing the number of subjects with olfactory & taste disturbances who have COVID-19 infection with the number of patients with olfactory & taste disturbances, and multiplying by 100%
Specificity of olfactory and taste disturbances in predicting COVID-19 infection | Baseline
  The percentage of true negatives, i.e. the proportion of patients without olfactory and taste disorders who do not have COVID-19 infection. This can be calculated by dividing the number of subjects without olfactory & taste disturbances who do not have COVID-19 infection with the number of patients without olfactory & taste disturbances, and multiplying by 100%

CONTACTS AND LOCATIONS:
Overall Officials: Siti Sabzah Mohd Hashim, MD MS, Study Chair — Hospital Sultanah Bahiyah
Locations (14):
- Malaysia (14):
  - Hospital Enche' Besar Hajjah Khalsom, Kluang, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Tuanku Jaafar, Seremban, Negeri Sembilan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Tuanku Fauziah, Kangar, Perlis
  - Penang Hospital, George Town, Pulau Pinang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
  - Kuala Lumpur General Hospital, Kuala Lumpur
  - Hospital Melaka, Malacca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Giacomelli A, Pezzati L, Conti F, Bernacchia D, Siano M, Oreni L, Rusconi S, Gervasoni C, Ridolfo AL, Rizzardini G, Antinori S, Galli M. Self-reported Olfactory and Taste Disorders in Patients With Severe Acute Respiratory Coronavirus 2 Infection: A Cross-sectional Study. Clin Infect Dis. 2020 Jul 28;71(15):889-890. doi: 10.1093/cid/ciaa330. No abstract available. PMID 32215618
- [Background] Mao L, Jin H, Wang M, Hu Y, Chen S, He Q, Chang J, Hong C, Zhou Y, Wang D, Miao X, Li Y, Hu B. Neurologic Manifestations of Hospitalized Patients With Coronavirus Disease 2019 in Wuhan, China. JAMA Neurol. 2020 Jun 1;77(6):683-690. doi: 10.1001/jamaneurol.2020.1127. PMID 32275288
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Kaye R, Chang CWD, Kazahaya K, Brereton J, Denneny JC 3rd. COVID-19 Anosmia Reporting Tool: Initial Findings. Otolaryngol Head Neck Surg. 2020 Jul;163(1):132-134. doi: 10.1177/0194599820922992. Epub 2020 Apr 28. PMID 32340555
- [Background] Yan CH, Faraji F, Prajapati DP, Boone CE, DeConde AS. Association of chemosensory dysfunction and COVID-19 in patients presenting with influenza-like symptoms. Int Forum Allergy Rhinol. 2020 Jul;10(7):806-813. doi: 10.1002/alr.22579. Epub 2020 Jun 1. PMID 32279441
- [Background] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008
- See also: AAO-HNS: Anosmia, Hyposmia, and Dysgeusia Symptoms of Coronavirus Disease | American Academy of Otolaryngology-Head and Neck Surgery — https://www.entnet.org/content/aao-hns-anosmia-hyposmia-and-dysgeusia-symptoms-coronavirus-disease